CLINICAL TRIAL: NCT00209469
Title: Double Blind Controlled Trial of Alendronate for the Treatment of Childhood and Adolescent Glucocorticoid-Associated Osteopenia and Osteoporosis
Brief Title: Network Osteoporosis Study
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glaser Pediatric Research Network (Network)
Collaborators: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GPRN1.OSTEO.PL.6.0
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Osteopenia; Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Alendronate

INTERVENTIONS:
Drug: alendronate sodium

SUMMARY:
This study is evaluating the use of the drug alendronate in preventing or reversing bone loss in children and adolescents receiving steroid medications.

DETAILED DESCRIPTION:
This trial will test the hypothesis that among 90 children and adolescents with Crohn's disease, ulcerative colitis, systemic-onset juvenile rheumatoid arthritis, juvenile dermatomyositis, systemic lupus erythematosus, mixed connective tissue disease and vasculitis, treatment of glucocorticoid-associated osteopenia and osteoporosis with 18 months of alendronate (FOSAMAX®, Merck & Co., Inc.) will result in greater improvement in the mean change of individual AP spine bone mineral density (BMD) (gm/cm2) determined by dual energy X-ray absorptiometry (DXA) than treatment with 18 months of standard of care therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be diagnosed with either ulcerative colitis, Crohn's disease, systemic-onset juvenile rheumatoid arthritis, juvenile dermatomyositis, systemic lupus erythematosus (SLE), mixed connective tissue disease (MCTD) or vasculitis according to standard criteria where available, and according to treating physicians when not available.
* Subjects must have diminished AP lumbar spine (L1-L4) BMD by DXA (Hologic 4500) with a Z score ≤ -1.5 SD assessed within 8 weeks of the Baseline Visit.
* Subjects must have received daily, alternate day or weekly systemic glucocorticoid therapy for a minimum of six months total in their life-time.
* Subjects must be between the ages of 8 and 21 years, 11 months, at randomization. Although subjects younger than 8 years of age may be affected by osteoporosis, limited normative data prevents assignment of a BMD Z score for this group. Subjects through 21 years, 11 months will be included because many individuals with chronic disorders will have an immature skeleton, and even in healthy individuals there is significant accrual of bone mass into the 20's, making this a dynamic and critical time period for analysis.
* Females who have had at least one menstrual cycle must either be abstinent or must be using an effective method of birth control (e.g. intrauterine contraceptive device, oral contraceptive, diaphragm or condom with contraceptive jelly, cream, or foam). This will be documented at each visit. Additionally, they must test negative on a urine pregnancy test which will be administered at every visit. Subjects will be informed that because the drug remains in the body for many years, it is possible that a developing fetus could be harmed by the drug even if a woman stops taking the drug long before she becomes pregnant.

Exclusion Criteria:

* Current or recent (within 6 months) treatment with therapeutic doses of a bisphosphonate, calcitonin, human growth hormone, and heparin, all agents known to alter bone density
* A history of recent (within one year of screening) major upper gastrointestinal (GI) disease (above the jejunum), including, but not limited to, peptic ulcer, esophageal disease or active GI bleeding, or ever had surgery of the upper GI tract other than pyloroplasty. A history of abnormalities of the esophagus which delay esophageal emptying, such as stricture or achalasia
* Hyperthyroidism (suppressed thyroid stimulating hormone (TSH) and elevated free thyroxine (T4)), hyperparathyroidism (elevated parathyroid hormone (PTH)), malignancy, rickets, or osteomalacia (by history), all assessed within 8 weeks of the Baseline Visit.
* 25 (OH) vitamin D below 20 g/L
* Planned or current pregnancy and/or breastfeeding
* Renal dysfunction defined as dependence on dialysis or a creatinine clearance < 35 ml/min, assessed within 4 weeks of the Baseline Visit. Creatinine clearance = [(height in cm x 0.55)/plasma creatinine] for all females and for males < 13 years old; [(height in cm x 0.70)/plasma creatinine] for males  13 years old.
* Hepatic insufficiency defined as SGPT or SGOT greater than twice normal for age, assessed within 4 weeks of the Baseline Visit.
* Uncorrected hypocalcemia (ionized calcium>10% below age-adjusted range), assessed within 4 weeks of the Baseline Visit.
* Known or suspected hypersensitivity to bisphosphonates
* Inability to follow instructions for dosing, including being unable to swallow the study medication with plain water first thing in the morning, stand or sit upright without any other food or beverage for at least 30 minutes following dosing and until their next meal
* Weight greater than 136 kg (300 lb), as the DXA is not reliable for subjects of this size
* Weight less than 17 kg (37 lb), assessed within 8 weeks of the Baseline Visit.
* Permanent foreign body (prosthetic, surgical clips, permanent earring/umbilical ring) in region of interest, or soft tissue calcinosis overlying the region of interest
* Inability to undergo dual energy X-ray absorptiometry or CT scan
* Developmental or cognitive delay which may interfere with cooperation and/or compliance with the procedures
* Subject expects to move out of the area during the study period, rendering follow-up per protocol impractical
* Subject has any other condition or therapy that, in the opinion of the investigator, might pose a risk to the subject or confound the results of the study.

Ages: 8 Years to 22 Years | Sex: All
Age Groups: Child, Adult
Enrollment: 90
Dates: Start 2002-07; Study Completion 2007-02

PRIMARY OUTCOMES:
Mean change of individual AP spine BMD (gm/cm2) determined by dual energy X-ray absorptiometry (DXA) at 6, 12,18, 24 and 30 Months.

CONTACTS AND LOCATIONS:
Overall Officials: Emily von Scheven, MD, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Children's Hospital, Boston, Boston, Massachusetts